CLINICAL TRIAL: NCT02384408
Title: Comparative Effects of Drospirenone and Tibolone on the Postmenopausal Endometrium
Brief Title: Hormone Replacement Therapy on the Postmenopausal Endometrium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Collaborators: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Benedito Fabiano dos Reis, Professor, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 10979112.1.3001.5479; 598.391-0 (Other: FCMSCSP)
Record Dates: First submitted 2015-02-03; First posted 2015-03-10 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Menopause
Keywords: menopause; drospirenone; tibolone; Bcl-2; steroid receptors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Control Group: Women without hormone replacement therapy. Transvaginal Ultrasound - Endometrial Thickness; Endometrial Biopsy. Endometrial Immunohistochemical Study
  Interventions: Procedure: Endometrial Biopsy; Device: Transvaginal Ultrasound; Procedure: Endometrial Immunohistochemical
- Hormone treatment (Experimental): Group Drospirenone: To whom a continuous combined treatment with drospirenone 2 mg and 17β-estradiol 1 mg (DRSP/E2) will be administered daily for 24 weeks.
  Group Tibolone: To whom treatment with tibolone 1.25 mg (Tib) will be administered daily for 24 weeks.
  Transvaginal Ultrasound - Endometrial Thickness; Endometrial Biopsy. Endometrial Immunohistochemical Study
  Interventions: Procedure: Endometrial Biopsy; Device: Transvaginal Ultrasound; Procedure: Endometrial Immunohistochemical

INTERVENTIONS:
Procedure: Endometrial Biopsy — Histological assessment
Device: Transvaginal Ultrasound — Endometrial Thickness made by ultrasound
  Other Names: Endometrial Thickness
Procedure: Endometrial Immunohistochemical — Immunoexpression of estrogen (ER) and progesterone receptors (PR) and Bcl-2 protein

SUMMARY:
Healthy postmenopausal women, amenorrheic for 1-10 years, aged 45-60 years and in use of follicle stimulating hormone > 30 mille-International unit/milliliters (mIU/mL), will participate in the study.

All women will be informed by a physician of the risks and possible benefits of Hormone Replacement Therapy (HRT).

The continuous combined treatment with drospirenone 2 mg and 17β-estradiol 1 mg or tibolone 1.25 mg will be administered for a 24-week period.

Transvaginal ultrasound was performed to evaluate the thickness of the endometrium at baseline. At study end-point, an endometrial biopsy will be performed with a Pipelle endometrial sampler to examine histological and immunohistochemical parameters.

Immunohistochemical detection of Bcl-2 protein, estrogen and progesterone receptors will be performed in stroma and glandular epithelium.

DETAILED DESCRIPTION:
Subjects

Healthy postmenopausal women, amenorrheic for 1-10 years, aged 45-60 years and in use of follicle stimulating hormone > 30 mille-International unit/milliliters (mIU/mL), will participate in the study.

All women will be informed about the trial and signed the informed consent documents, eligibility was determined based on medical history, and on general physical and gynecological examination. All women were informed by a physician of the risks and possible benefits of Hormone Replacement Therapy (HRT). Upon inclusion, Transvaginal ultrasound (TV-US) was performed to evaluate the thickness of the endometrium at baseline. At study end-point, an endometrial biopsy will be performed with a Pipelle endometrial sampler to examine histological and immunohistochemical parameters . Vital signs, blood pressure, weight, Pap smear, mammography, routine clinical chemistry assays (including, cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol, triglycerides) and hematology will also be evaluated at screening.

Treatment Groups Of the 100 women initially evaluated, 32 did not meet the inclusion and exclusion criteria, while eight refused to participate, giving a final total of 60 patients for inclusion in the study. The sixty postmenopausal women were randomly allocated into three groups: Group I: control group comprising 20 patients (no hormonal treatment); Group II: also comprising 20 patients, to whom a continuous combined treatment with drospirenone 2 mg and 17β-estradiol 1 mg (DRSP/E2) will be administered daily; and Group III: also comprising 20 patients, to whom treatment with tibolone 1.25 mg (Tib) will be administered daily. All treatments will be administered for a 24-week period. DRSP/E2 was purchased from "Bayer Schering Pharma™", Brazil and Tib from "Biolab™", Brazil. The duration of the treatment will be 6 cycles, each lasting a period of 28 days (conducted for a total of 24 weeks). Randomization will be done with the aid of computer software in order to prevent bias in the selection process.

Objective: A prospective randomized controlled trial will be conducted to evaluate the effect of low dose of tibolone and estradiol/drospirenone on the histology, expression of estrogen (ER) and progesterone receptors (PR) and Bcl-2 protein, in endometrium of postmenopausal women.

The effects on endometrial thickness will be determined by Transvaginal Ultrasound (TV-USG) at study baseline and again after 6 cycles of treatment in all women participants. Scans were performed with a real-time scanner, "Hitachi 405"ultrasound system equipped with a 5.0-megahertz (MHz) vaginal transducer, at the "Vale do Sapucai University". An endometrial thickness < 4 millimeters (mm) will be interpreted as not supporting a diagnosis of endometrial cancer.

Endometrial biopsy and sampling will be performed at the end of the treatment course using a "Pipelle Curette" de Cornier, placed high into the upper fundus of the uterus. An aliquot of the endometrial sample will be pushed from the pipette into a polypropylene vial. The vial will be capped, immediately frozen, and then stored at -20º Celsius until shipping in dry ice to the Department of Pathology at the "Vale do Sapucai University", directed by one of the authors, for measurement of Progestogen Receptor (PR) and Estrogen Receptor (ER) receptors as well as Bcl-2 protein. The remaining endometrial tissue will fix in 10% neutral buffered formalin for 6-48 h and then process into paraffin blocks.

Histological and immunohistochemical assessment Histology classification will be carried out by two pathologists. Both pathologists will do a blind reading of different tissue sections of the same block-sample. After staining with hematoxylin/eosin and Schiff Periodic Acid (PAS), each specimen was classified into one of the following categories: tissue insufficient for diagnosis, atrophic and/or inactive endometrium, proliferative or weakly proliferative endometrium, and progestogenic .

Immunohistochemical detection of Bcl-2 protein will be performed by two pathologists. After antigen retrieval and blocking of non-specific sites with normal serum using the Avidin/Biotin Blocking kit (Vector Laboratories, Inc, California, USA), the sections will be incubated overnight at 4º Celsius with anti-Bcl-2 mouse monoclonal antibody (1:100, Clone 124, DAKO, Denmark). The tissue-bound antibody will be incubated for 30 min at room temperature with the Envision System. Staining will be visualized by use of Envision (Kit N1587, DAKO, Denmark). The cellular staining pattern for this antibody is cytoplasmic. The presence of ER and PR will be detected as described previously. The cellular staining patterns for these antibodies are nuclear. A breast cancer specimen will be used as a positive control for the steroid receptors.

Examinations and photography will performed using an "Axioskop 40 - Zeiss" light microscope equipped with a Canon™ D30 digital camera (Tokyo, Japan) and video monitor (LG 14" LCD) according to the procedures of the Pathology Department from Santa Casa of Sao Paulo Medical School, Sao Paulo, Brazil.

The morphometric technique for immunohistochemistry quantification will be done with the aid of a Neubauer graduated chamber. This consists of a glass slide, thicker than a regular slide, each having a grid design dividing it into squares with known dimensions, visualized only through an optical microscope. The Neubauer counting chamber is divided into 9 large squares, each with 1 mm sides, by means of triple lines (thus area of a large square= 1 mm²). Each large square contains 16 (4 x 4) medium-size squares. Each medium size square is further divided by triple lines into 25 (5 x 5) smaller squares, each with a side length of 1/5 of a mm. Thus, the area of an individual small square is 0.05 x 0.05 mm= 0.0025 mm² and 0.1 mm deep .

The image observed through the microscope lenses will be captured by the video camera and displayed on the chosen monitor. The Neubauer chamber will be then placed under the optical microscope, using an objective which magnifies the original size of the object by 400x or by any other magnification elected by the researcher. Finally, the area under the high magnification field (400x magnification) is estimated in mm² by counting the total number of individual small 0.0025 mm² squares of the chamber within the magnification area chosen. The total area under high magnification corresponded to 0.094 mm².

Using this approach, each section prepared by the immunohistochemical method will be evaluated under the light microscope. The number of cells in the study will be counted at 400x magnification. A 10-field count will be performed in the different situations evaluated. The mean number of cells present in this 10-field count represented an area of 0.094 mm². By means of a simple rule of three, the number of cells will be converted into 1 mm² counts. The cell count will be expressed as numerical density, i.e. number of positive cells per square millimeter of epithelium.

The number of Bcl-2-positive cells and immunoreactivity for PR and ER expression will quantified manually by two trained observers, blind to the experiment, and will evaluate separately for glandular and stromal cells. The immunohistochemical staining index (numerical density) will be defined as the mean number of positive immunoexpression cells per mm², calculate in 10 different fields.

Statistical analysis Statistical analysis will be performed using the "StatistiXL Package™" (Statistical Power for Microsoft Excel version 1.8, 2007). Differences in demographic parameters, immunohistochemical staining index of ER, PR and Bcl-2 protein expression (numerical density), as well as baseline and treatment end-point endometrial thickness, will be analyzed by the paired Student's t-test in the different groups. The relationships between ER, PR and Bcl-2 protein expression in stroma and glandular epithelium will be analyzed using Spearman's test.

Statistical significance will set at p < 0.05. Data will express as mean + standard deviation (SD).

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women, amenorrheic for 1-10 years,
* aged 45-60 years and in use of follicle stimulating hormone > 30 mIU/mL, participated in the study.
* In all subjects, menopausal status will be confirmed by levels of serum follicle stimulating hormone and estradiol in the postmenopausal range.

Inclusion criteria will be:

* an intact uterus,
* a washout period of 8 weeks for oral estrogens with or without progestogens, androgens, or selective estrogen receptor modulators (SERMs), four weeks for transdermal or local sex steroids, and 20 weeks for injections of medroxyprogesterone acetate (MPA) containing contraceptives.

Exclusion Criteria:

* neoplastic, metabolic and infectious diseases,
* a uterine size greater than that consistent with a 12-week gestation,
* any abnormality on bimanual pelvic examination,
* concomitant use of any hormonal drug,
* body mass index (BMI) > 30 kg/m2,
* cigarette smoking and an endometrial thickness > 5 mm or the presence of any endometrial abnormalities on transvaginal ultrasound (TV-US).
* No subjects have present or past history of venous thrombosis, cerebrovascular or cardiovascular disease, and
* women were excluded if they had any condition that could alter the pharmacokinetics or hypersensitivity to drospirenone/estradiol and tibolone.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The endometrium thickness | up to 24 weeks
  Transvaginal ultrasound will be performed to evaluate the thickness of the endometrium in milimiters at baseline and the end of the study in postmenopausal women under use of drospirenone and tibolone. The results will be expressed as mean and standard deviation.

SECONDARY OUTCOMES:
Bcl-2 protein in postmenopausal endometrium | 24 weeks
  Histological and immunohistochemical detection of Bcl-2 protein will be performed on postmenopausal endometrium. The cell count will be expressed as numerical density, i.e. number of positive cells per square millimeter of epithelium.
Estrogen and progestogen receptors in postmenopausal endometrium | 24 weeks
  The presence of estrogen and progestogen receptors will be performed on postmenopausal endometrium. The cell count will be expressed as numerical density, i.e. number of positive cells per square millimeter of epithelium.

CONTACTS AND LOCATIONS:
Overall Officials: Benedito F Reis, Prof, Principal Investigator — Faculdade de Ciências Médicas da Santa Casa de São Paulo
Locations (1):
- Vale Do Sapucai University (Univas), Pouso Alegre, Minas Gerais, Brazil

REFERENCES:
- [Result] Klaassens AH, van Wijk FH, Hanifi-Moghaddam P, Sijmons B, Ewing PC, Ten Kate-Booij MJ, Kooi GS, Kloosterboer HJ, Blok LJ, Burger CW. Histological and immunohistochemical evaluation of postmenopausal endometrium after 3 weeks of treatment with tibolone, estrogen only, or estrogen plus progestagen. Fertil Steril. 2006 Aug;86(2):352-61. doi: 10.1016/j.fertnstert.2005.12.077. Epub 2006 Jul 7. PMID 16828477
- [Result] Lima SM, Reis BF, Yamada SS, Postigo S, Grande RM, Botogoski SR, Campaner AB, Hueb CK, Galvao MA. Effects of drospirenone/estradiol on steroid receptors and Bcl-2 in the postmenopausal endometrium. Climacteric. 2011 Oct;14(5):551-7. doi: 10.3109/13697137.2011.559604. Epub 2011 Apr 6. PMID 21469974
- [Result] Campaner AB, Longo Galvao MA. Application of an easy and useful morphometric technique for immunohistochemistry counting. Gynecol Oncol. 2009 Jan;112(1):282-3. doi: 10.1016/j.ygyno.2008.08.012. Epub 2008 Oct 19. No abstract available. PMID 18937967
- [Result] Kloosterboer HJ. Tissue-selectivity: the mechanism of action of tibolone. Maturitas. 2004 Aug 30;48 Suppl 1:S30-40. doi: 10.1016/j.maturitas.2004.02.012. PMID 15337246
- [Result] Grady D, Gebretsadik T, Kerlikowske K, Ernster V, Petitti D. Hormone replacement therapy and endometrial cancer risk: a meta-analysis. Obstet Gynecol. 1995 Feb;85(2):304-13. doi: 10.1016/0029-7844(94)00383-O. PMID 7824251
- [Result] Smith-Bindman R, Kerlikowske K, Feldstein VA, Subak L, Scheidler J, Segal M, Brand R, Grady D. Endovaginal ultrasound to exclude endometrial cancer and other endometrial abnormalities. JAMA. 1998 Nov 4;280(17):1510-7. doi: 10.1001/jama.280.17.1510. PMID 9809732
- [Result] Gokaslan H, Oktem O, Durmusoglu F, Eren F. Apoptosis in the endometrium of postmenopausal women receiving tibolone. Gynecol Obstet Invest. 2003;56(3):124-7. doi: 10.1159/000073624. Epub 2003 Sep 22. PMID 14504425